CLINICAL TRIAL: NCT05377411
Title: SMART Stimulation: Precision Neuromodulation of Cognition in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Soterix Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB202100953
Record Dates: First submitted 2022-04-07; First posted 2022-05-17 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-10

CONDITIONS: Aging
Keywords: tdcs; cognitive training
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Intervention Model Description: Arm 1 will receive optimized tDCS paired with cognitive training. Arm 2 will receive sham tDCS paired with cognitive training.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Procedures for tDCS will be identical for both arms with the exception of the amount of current delivered. Neither the participant nor the experimenter will know the amount of current delivered during tDCS sessions. Web-based permuted block randomization to randomly divide participants into the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Optimized tDCS + Cognitive Training (Experimental): A Soterix Clinical Trials Direct Current Stimulator will apply 20 minutes of up to 4.0mA direct current through two biocarbon rubber electrodes covered with at least 5mm-thick conductive electrode paste buffer, and placed over the optimized locations based on the international 10-20 system by using a combination of 10-20 EEG cap measurement and a stereotactic neuronavigation system. Stereotactic neuronavigation will be used as needed and may not be used on all participants.
  Interventions: Device: tDCS; Behavioral: cognitive training
- Sham tDCS + Cognitive Training (Sham Comparator): Sham stimulation is performed with the same device and all procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of up to 4 mA of direct current stimulation at the beginning of the session. Participants habituate to the sensation of tDCS within 30-60 seconds of stimulation. This procedure provides the same sensation of tDCS without the full duration of stimulation, making it a highly effective sham procedure.
  Interventions: Device: tDCS; Behavioral: cognitive training

INTERVENTIONS:
Device: tDCS — During tDCS, a weak electrical current is applied to the scalp that penetrates skin, bone, CSF and the meninges to stimulate underlying cortical and subcortical tissue
Behavioral: cognitive training — Cognitive Training (CT) will involve up to 10 hours of training over 2-weeks (10 days). CT employs a PositScience BrainHQ suite via its researcher portal. These tasks are web-based and multi-platform (i.e., Windows, Mac). Participants will be randomly assigned to training on 4 tasks focusing on working memory or 4 tasks focusing on attention/speed of processing.

SUMMARY:
The current study will investigate methods for enhancing cognitive training (CT) effects in healthy older adults by employing a combination of interventions facilitating neural plasticity and optimizing readiness for learning. A pilot randomized clinical trial will examine the individual and combined impact of pairing cognitive training with transcranial direct current stimulation (tDCS). A precision dosing algorithm will be used to determine the appropriate levels of current and location of electrodes to deliver current using tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age: 65 to 89 years
* English speaking
* Physically mobile
* Working memory function between 0-75th percentile determined by screening results on the POSIT Baseline Cognitive Training computerized tasks.

Exclusion Criteria:

* Neurological disorders (e.g., dementia, stroke, seizures, traumatic brain injury).
* Evidence of dementia (NACC UDS scores of 1.5 standard deviations below the mean for age, sex and education adjusted norms in a single cognitive domain on the task).
* Past opportunistic brain infection
* Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis or severe major depression and/or suicidality.
* Unstable (e.g., cancer other than basal cell skin) and chronic (e.g, severe diabetes) medical conditions.
* MRI contraindications (e.g., pregnancy, claustrophobia, metal implants that are contraindicated for MRI).
* Physical impairment precluding motor response or lying still for 1 hr and inability to walk two blocks without stopping.
* Certain prescription medications may possibly reduce effects otherwise induced by the tDCS stimulation protocol.
* Hearing or vision deficits that will not allow for standardized cognitive training stimulation; ie colorblindness, inability to hear through headphones (with or without hearing aids), macular degeneration or other significant diseases that cause severe loss of vision. If vision is corrected with lenses to appropriate levels, then participant will be eligible.
* Left handedness, as those with left-handedness have a higher percentage rate of atypical functional lateralization for brain functions, which would significantly interfere with interpretability of brain data.
* Participants with precision tDCS dosage of >4.0mA required will be excluded due to limitations of tDCS device (maximum output of 4.0 mA). The maximum output of 4.0 mA reflects a technical limitation of the device design rather than a safety threshold.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McKnight Brain Institute, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optimized tDCS + Cognitive Training | Sham tDCS + Cognitive Training
Started | 17 | 16
Completed | 16 | 15
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimized tDCS + Cognitive Training | Sham tDCS + Cognitive Training | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.65 (5.31) | 72.25 (5.86) | 72.45 (5.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 15 | 30
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: N-Back Working Memory
Description: Change in working memory performance on the N back working memory MRI task from baseline to post test will be assessed. Post test will occur approximately two weeks following baseline.
  The N-back working memory task will be completed during the MRI scan at both baseline and post test assessments. Working memory performance will be defined as a composite of reaction time and accuracy for two back trials. Specifically Target Accuracy percent correct and average correct target reaction time in milliseconds. Percent changes were calculated for Target Accuracy and Reaction Time in the form of (post test-pre test)/pre test. Since the direction of improvement is opposite for the two variables (i.e. higher Accuracy is better and lower Reaction Time is better), the reaction time percent change was multiplied by -1 to ensure a larger number indicated improved performance. To create a composite these two percent changes (Target Accuracy and Reaction Time) were averaged into a single value.
Time Frame: Baseline to post test. Post test will occur approximately two weeks following baseline.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Optimized tDCS + Cognitive Training | Sham tDCS + Cognitive Training
Number analyzed (Participants) | 16 | 15
percent change | .2030 (.3164) | .0731 (.1404)

ADVERSE EVENTS:
Time Frame: 2 weeks. Adverse events were collected from study enrollment (week 0) until post-test (week 2).
Description: Adverse events were collected at baseline and post-test assessments via medical questionnaires. Adverse events could be reported outside of baseline and post-test assessments via participant self-reporting to experimenters during the approximate two week period of intervention.
Arm/Group | Optimized tDCS + Cognitive Training | Sham tDCS + Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 7/17 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optimized tDCS + Cognitive Training (N=17) | Sham tDCS + Cognitive Training (N=16)
Headache (General disorders) | 4 | 3
Eye Redness (Eye disorders) | 1 | 1
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Car accident (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT05377411/Prot_SAP_000.pdf